CLINICAL TRIAL: NCT04056754
Title: A Randomised, Double-Blind, Multicentre Phase Ⅲ Study to Evaluate Abiraterone Acetate Versus Placebo Combined With Prednisone in Subjects With Asymptomatic or Mild Symptoms Without Chemotherapy, Metastatic Castration Resistant Prostate Cancer.
Brief Title: Study of Abiraterone Acetate in Subjects With Metastatic Castration Resistant Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTTQL-ABTL
Record Dates: First submitted 2019-08-11; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2016-04

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
MeSH Terms: interventions — Abiraterone Acetate; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abiraterone acetate group (Experimental): Subjects in this group administered 4 tablets abiraterone acetate once daily and 5mg prednisone twice daily, in 28-day cycle on fasting conditions.
  Interventions: Drug: Abiraterone Acetate; Drug: Prednisone
- Placebo group (Placebo Comparator): Subjects in this group administered 4 tablets abiraterone acetate blank analog tablet once daily and 5mg prednisone twice daily, in 28-day cycle on fasting conditions.
  Interventions: Drug: Placebo; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone Acetate — Subjects administered 4 tablets abiraterone acetate twice daily in 28-day cycle.
  Arms: Abiraterone acetate group
Drug: Placebo — Subjects administered 4 tablets abiraterone acetate blank analog tablet twice daily in 28-day cycle.
  Arms: Placebo group
Drug: Prednisone — Subjects administered 5mg prednisone twice daily in 28-day cycle.

SUMMARY:
Abiraterone acetate is an orally effective CYP17 inhibitor, which is metabolized into abiraterone in the body, and its inhibitory activity against CYP17 is 10-30 times that of ketoconazole. Clinical studies have shown that abiraterone acetate can significantly reduce the level of prostate specific antigen (PSA) in PCa patients, and help to reduce tumors, extending the lifespan of patients with advanced PCa for several years, and the toxicity is acceptable.

ELIGIBILITY:
Inclusion Criteria:

- 1.18 years and older, Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1, Life expectancy ≥ 6 months.

2. Prostate cancer. 3. Serum testosterone <50 ng/dL (or 1.7 nmol/L). 4. Prostate cancer progression or lesion metastasis. 5. Restriction of antiandrogen therapy. 6. Restriction of Radiation therapy. 7. The treatment period of ketoconazole for prostate cancer was not exceed 7 days.

8. Has not used opioid analgesics and azole drugs within 4 weeks before the first dose.

9. Question 3 of the Concise Pain Questionnaire (BPI-SF) scored from 0-3 points.

10. Adequate laboratory indicators. 11. Must be able to swallow tablets. 12. No pregnant or breastfeeding women, and a negative pregnancy test. 13. Understood and signed an informed consent form.

Exclusion Criteria:

1. Prostate pathology results are neuroendocrine prostate cancer.
2. Has received cytotoxic chemotherapy or biological therapy for metastatic castration resistant prostate cancer.
3. Has contraindications to the use of prednisone.
4. A chronic disease that exceeds the prednisone dose in the study.
5. Uncontrolled high blood pressure.
6. Active or symptomatic viral hepatitis or other chronic liver disease.
7. Visceral metastasis or brain metastasis.
8. Pituitary or adrenal dysfunction.
9. Active autoimmune diseases require the use of hormone therapy.
10. Clinically significant heart disease.
11. Participated in other clinical trials within 4 weeks.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2014-07-16 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Time to PSA progression (TTPP） | Baseline up to 24 months
  The time interval between the administration of the drug and the progression of serum prostate specific antigen (PSA).

SECONDARY OUTCOMES:
Prostate specific antigen remission time | Baseline up to 24 months
  It was ≥50% lower than the baseline, and was confirmed as remission after re-testing after ≥4 weeks.
Objective Response Rate (ORR) | Baseline up to 24 months
  The percentage of participants with a best overall response defined as complete response (CR) or partial response (PR).
Eastern Cooperative Oncology Group (ECOG) | Baseline up to 24 months
  The ECOG scoring standard is an indicator of the general health status and tolerance to treatment from the patient's physical strength. ECOG physical status score standard from 0 to 5. Starting with the dose until the score increases from the baseline.
Overall Survival (OS) | Baseline up to 24 months
  Time from date of randomization to date of death due to any cause.
To pain progression time | Baseline up to 24 months
  Time from the start of medication to the progression of pain.
Quality of life assessment scale (FACT-P) | Baseline up to 24 months
  Functional Assessment of Cancer Therapy- Prostate Cancer (FACT-P) total score, Functional Assessment of Cancer Therapy- General (FACT-G) total score, trial outcome index, functional well-being, physical well-being, prostate cancer subscale, and Functional Assessment of Cancer Therapy (FACT) Advanced Prostate Symptom Index-6 (FAPSI-6).
Prostate specific antigen remission rate | Baseline up to 24 months
  The remission rate was defined as the proportion of remissions to the total number of people.

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Sun-Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Guangzhou Military Region Wuhan General Hospital, Wuhan, Hubei
  - TongJi medical college of HuaZhong University of Science & Technology Affiliated TongJi Hospital, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Fudan University Medical College Affiliated Huadong Hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - RenJi Hospital of Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital of Zhenjiang University School of Medicine, Hangzhou, Zhejiang